CLINICAL TRIAL: NCT05782101
Title: Integrated Proteomic HPLC-ESI-MS Analysis of Salivary Peptides of Preterm Newborns: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4242
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Bronchopulmonary Dysplasia; Retinopathy of Prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bronchopulmonary Dysplasia/Retinopathy of prematurity: Preterm neonates whith Bronchopulmonary dysplasia and/or Retinopathy of prematurity
  Interventions: Diagnostic Test: Integrated proteomic HPLC-ESI-MS analysis of salivary peptides
- No Bronchopulmonary Dysplasia/Retinopathy of prematurity: Preterm neonates without Bronchopulmonary Dysplasia and/or Retinopathy of prematurity
  Interventions: Diagnostic Test: Integrated proteomic HPLC-ESI-MS analysis of salivary peptides

INTERVENTIONS:
Diagnostic Test: Integrated proteomic HPLC-ESI-MS analysis of salivary peptides — A targeted ESI mass spectrometry investigation, based on a top-down analysis of the intact salivary proteome will be performed.

SUMMARY:
The analysis of saliva of preterm newborns could be a powerful tool to investigate human fetal development in an ethically acceptable fashion, indeed the collection of salivary samples is a fast and non-invasive procedure. The purpose of the study is to characterize peptide and proteins present in human preterm saliva and to investigate the relative amount of several proteoforms of the proteins and peptides detectable in preterm saliva in order to have information on the activity of various enzymes acting during late fetal development. Preterm infants with gestational age between 175-216 days (25-30 weeks), admitted to the Neonatal Intensive Care Unit (NICU) will be enrolled for this study. A saliva sample will be collected every seven days from the birthday and up to 40 weeks (286 days) of postmenstrual age (PMA) or up to discharge if it occurs earlier. A targeted ESI mass spectrometry investigation, based on a top-down analysis of the intact salivary proteome will be performed.

DETAILED DESCRIPTION:
Background

The study of human fetal development is hampered by the difficulty to have an experimental plan and a specimen collection ethically acceptable. In the past years the analysis of saliva of preterm newborns is demonstrated to be a powerful tool to investigate human fetal development in an ethically acceptable fashion [1]. The collection of salivary samples is indeed a non-invasive procedure which is usually performed by the personnel of the Neonatology Unity for the wellbeing and survival of highly preterm newborns. The samples collected are usually discharged, while their analysis, after the informed consent of one of the parents, could be precious to investigate molecular events occurring during the last months of fetal life.

Indeed, previous HPLC-ESI-MS analyses carried out on salivary samples collected from newborns at different postmenstrual age (PMA) evidenced the presence of high levels of more than 40 proteins, many of them pertaining to the family of S100 proteins, decreasing their amounts according to the PMA [1]. Commonly, these proteins are either absent or present at a concentration near to the limit of sensitivity of our MS apparatus at the normal term of delivery and in adult saliva. In the first years of life these proteins are slowly replaced by the protein present in the human adult saliva [2]. The first adult salivary proteins appearing in the preterm newborn at 180-190 days of PMA are the acidic proline-rich proteins (aPRPs) isoforms encoded by the PRH2 locus, together with a glycosylated basic proline-rich protein expressed by the PRB3 locus, followed at 210-220 days of PCA by histatins, statherin, and P-B peptide. Acidic proline-rich proteins encoded by PRH1 locus appeared in whole saliva of babies from 1 to 3 weeks after the normal term of delivery, S-type cystatins appeared at 1 year (±3 months), and basic proline-rich proteins appeared after 4 years (±1 year) of age and reach the level observed in the adult after the puberty [2]. These protein families specific of human adult saliva are differently secreted by the major salivary glands (parotid, submandibular and sublingual) and during the secretion process are submitted to several post-translational modifications (PTMs) under the action of various enzymes (i.e kinases and proteinases) common to other exocrine and endocrine organs [3-6]. Studies carried out by our research group showed for instance that the activity of Fam20C, a pleitropic Golgi kinase involved in the phosphorylation of many different substrates in many organs and tissues [7], responsible for the phosphorylation of aPRPs, histatin 1, statherin and S-type (salivary) cystatins is not active at 180 days of PMA. It slowly increases its activity reaching values comparable to adults at about 2 years of age [2,8]. Instead, MAPK14 involved in the phosphorylation of S100A9 was fully active since birth also in preterm newborns of 180 days of PMA [2]. These studies suggested also that the proteinases involved in the proteolysis of salivary proteins were more active in preterm newborns.

Aim of the study

The aim of the study will be to establish the structure and the relative amount over time of several peptides and proteins detectable in preterm saliva still pending for a precise characterization, with particular regard to enzymes with proteolytic or oxidative activity. Oxidative stress and proteolysis are well known pathogenetic mechanisms involved in pathological conditions of preterm infants such as bronchopulmonary dysplasia and retinopathy of prematurity [9-11]. A correlation of the different expression over time of the enzymes identified with the prevalence of these pathological conditions can be also evaluated and represent the basis for future studies aim to verify the utility of such peptides as pathological markers. The proteomic approach utilized will be a targeted ESI mass spectrometry, based on a top-down platform devoted to the analysis of the intact salivary proteome.

Materials and Methods

Setting The enrollment of newborns and the collection of saliva samples will be performed at the Complex Operative Unit of Neonatology of the Fondazione Policlinico Universitario A. Gemelli IRCCS of Rome. The treatment and proteomic analysis of the collected saliva samples will be performed at the Department of basic biotechnological, intensive and perioperative cares sciences of the Catholic University of the Sacred Heart of Rome.

The Proteomics and Metabolomics Unit of IRCCS-Fondazione Santa Lucia of Rome, the Department of Life and Environmental Sciences and Section of Pathological Anatomy of the Department of Medical Sciences and Public Health of Cagliary University and the "Giulio Natta" Institute of Chemical Sciences and Technologies - National Research Council, will contribute to the analysis of saliva samples and to data processing.

Study population and inclusion criteria The study will be carried out in accordance with the ethical standards laid down in the 1964 Declaration of Helsinki. All rules will be observed, and written consent forms will be signed by the donor or by parents of each child. For ethical reasons, saliva will be collected only when sample collection will cause no stress.

Preterm infants with gestational age between 175-216 days (25-30 weeks), admitted to the Neonatal Intensive Care Unit (NICU) will be enrolled for this study. Saliva sample will be collected at least even seven days from the birth date and up to 40 weeks (286 days) of PMA or up to discharge if it occurs earlier. Infants with major congenital malformations or prenatal infections will be excluded from the study.

As this is a pilot study, in the "pre-discovery" phase of characterization of the peptides, the calculation of the sample size is precluded.

However, it is possible to estimate the number of patients who can be enrolled in an appropriate timeframe: considering that in 2020, 75 newborns with gestational age between 25 and 30 weeks were hospitalized in the Neonatal Intensive Care Unit and among these 13 (17,3%) died, it can be estimated the possibility of studying at least 30 infants over a period of approximately 18 months.

The number of infants we intend to study is in line with the literature evidence for a pilot study [12].

Sample Collection and Treatment Whole saliva will be collected with a soft plastic aspirator as it flowed into the anterior floor of the mouth. After collection, each salivary sample will be immediately diluted 1:1 (v/v) with 0.2% aqueous 2,2,2-trifluoroacetic acid (TFA) on ice bath. The solution will be then centrifuged at 8000g for 5 min (4°C). Finally, the acidic supernatant will be separated from the pellet and either immediately analyzed with the HPLC-ESI-MS apparatus or stored at -80 °C until the analysis.

RP-HPLC-ESI-MS Analysis For low-resolution (1/6000) MS experiments the HPLC-ESI-IT-MS apparatus will be a Surveyor HPLC system (ThermoFisher Scientific) connected by a T splitter to a photo diode-array detector and either to an LCQ Advantage ion trap mass spectrometer (ThermoFisher Scientific).

High resolution analysis will be performed using a Nano-HPLC-nanoESI-Orbitrap Elite instrument. (Thermo Fisher Scientific). The injection volume will be 5 μL corresponding to 1 μg of total protein content per sample.

MS Analysis Deconvolution of low resolution averaged ESI-MS and ESI-MS/MS spectra will be automatically performed the HPLC-MS apparatus management software (Xcalibur 2.0.7 SP1, Thermo Fisher Scientific).

MS and MS/MS data obtained from bottom-up analyses will be elaborated by Proteome Discoverer 2.4 software (Thermo Fisher Scientific), based on the SEQUEST HT cluster as search engine against the Swiss-Prot Homo Sapiens proteome (UniProtKb, Swiss-Prot, Homo Sapiens).

Intact Protein/Peptide Characterization and Relative Quantification The different salivary proteins and their proteoforms investigated will be characterized by means of an integrated proteomic platform. [1] Salivary peptide and protein quantitative analysis of the saliva specimens will be based on the measurement of the low resolution HPLC-ESI-MS eXtracted Ion Current (XIC) peak area (signal/noise ratio >5). The XIC search reveals the peak associated with the protein of interest by extracting along the total ion current (TIC) chromatographic profile the intensity of the ion current of specific multiply charged ions (m/z) generated by the ESI source. The ions used to quantify the proteins and peptides will be chosen roughly in a number proportional to the protein mass and carefully selected to exclude values in common with other co-eluting peptides. The area of the XIC peak is proportional to protein/peptide concentration; therefore, under constant analytical conditions, it can be used for a quantitative analysis and comparative studies [13-14]. The estimated percentage error of the XIC procedure is <10%.

Statistical Analysis The characterization of the saliva in terms of peptides and proteins will be described with means and standard deviations for quantitative parameters. How the characterization changes over time (from the birthday - to 40 weeks) will be tested and any significant differences will be assessed through analysis of variance for repeated measures.

References

1. M. Castagnola, R. Inzitari, C. Fanali, F. Iavarone, A. Vitali, C. Desiderio, G. Vento, C. Tirone, C. Romagnoli, T. Cabras, B. Manconi, M.T. Sanna, R. Boi, E. Pisano, A. Olianas, M. Pellegrini, S. Nemolato, C.W. Heizmann, G. Faa, I. Messana. The surprising composition of the salivary proteome of preterm human newborn. Mol. Cell. Proteomics 10 (2011) M110.003467.
2. Messana I, Cabras T, Iavarone F, Manconi B, Huang L, Martelli C, Olianas A, Sanna MT, Pisano E, Sanna M, Arba M, D'Alessandro A, Desiderio C, Vitali A, Pirolli D, Tirone C, Lio A, Vento G, Romagnoli C, Cordaro M, Manni A, Gallenzi P, Fiorita A, Scarano E, Calò L, Passali GC, Picciotti PM, Paludetti G, Fanos V, Faa G, Castagnola M. Chrono-proteomics of human saliva: variations of the salivary proteome during human development. J Proteome Res. 14(4) (2015) 1666-1677.
3. Castagnola M., Cabras T., Vitali A., Sanna M.T., Messana I. Biotechnological implication of the salivary proteome. Trends Biotechnol. 29 (2011) 409-418.
4. I. Messana, T. Cabras, E. Pisano, M. T. Sanna, A. Olianas, B. Manconi, M. Pellegrini, G. Paludetti, E. Scarano, A. Fiorita, S. Agostino, A. M. Contucci, L. Calò, P. M. Picciotti, A. Manni, A. Bennick, A. Vitali, C. Fanali, R. Inzitari, M. Castagnola. Trafficking and post-secretory events responsible for the formation of secreted human salivary peptides. A proteomic approach. Mol. & Cell. Proteomics, 7 (2008) 911-926.
5. I. Messana, R. Inzitari, C. Fanali, T. Cabras, M. Castagnola. Facts and artifacts in proteomics of body fluids. What proteomics of saliva is telling us? J. Sep. Sci. 31 (2008) 1948-1963.
6. Castagnola, M.; Cabras, T.; Iavarone, F.; Vincenzoni, F.; Vitali, A.; Pisano, E.; Nemolato, S.; Scarano, E.; Fiorita, A.; Vento, G.; Tirone, C.; Romagnoli, C.; Cordaro, M.; Paludetti, G.; Faa, G.; Messana, I. Top-down platform for deciphering the human salivary proteome. J. Matern. Fetal Neonatal Med. 2012, 25 (Suppl 5), 27-43.
7. Tagliabracci VS, Wiley SE, Guo X, Kinch LN, Durrant E, Wen J, Xiao J, Cui J, Nguyen KB, Engel JL, Coon JJ, Grishin N, Pinna LA, Pagliarini DJ, Dixon JE. A Single Kinase Generates the Majority of the Secreted Phosphoproteome. Cell. 2015, 161(7):1619-32.
8. R. Inzitari, G. Vento, E. Capoluongo, S. Boccacci, C. Fanali, T. Cabras, C. Romagnoli, B. Giardina, I. Messana, M. Castagnola. Proteomic analysis of salivary acidic proline-rich proteins in human pre-term and at-term newborns. J. Proteome Res. 6 (2007) 1371-1377.
9. Capasso L, Vento G, Loddo C, Tirone C, Iavarone F, Raimondi F, Dani C, Fanos V. Oxidative Stress and Bronchopulmonary Dysplasia: Evidences From Microbiomics, Metabolomics, and Proteomics. Front Pediatr. 2019, 13;7:30. doi: 10.3389/fped.2019.00030.
10. Tirone C, Iavarone F, Tana M, Lio A, Aurilia C, Costa S, Castagnola M, Messana I, Vento G. Oxidative and Proteolytic Inactivation of Alpha-1 Antitrypsin in Bronchopulmonary Dysplasia Pathogenesis: A Top-Down Proteomic Bronchoalveolar Lavage Fluid Analysis. Front Pediatr. 2021, 23;9:597415. doi: 10.3389/fped.2021.597415.
11. Graziosi A, Perrotta M, Russo D, Gasparroni G, D'Egidio C, Marinelli B, Di Marzio G, Falconio G, Mastropasqua L, Li Volti G, Mangifesta R, Gazzolo D. Oxidative Stress Markers and the Retinopathy of Prematurity. J Clin Med. 2020 Aug 21;9(9):2711. doi: 10.3390/jcm9092711.
12. Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceut. Statist. 2005; 4: 287-291. DOI: 10.1002/pst.185
13. Levin, Y.; Schwarz, E.; Wang, L.; Leweke, F. M.; Bahn, S. Labelfree LC-MS/MS quantitative proteomics for large-scale biomarker discovery in complex samples. J. Sep. Sci. 2007, 30, 2198-2203.
14. Ong, S. E.; Mann, M. Mass spectrometry-based proteomics turns quantitative. Nat. Chem. Biol. 2005, 1, 252-262.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age between 175-216 days (25-30 weeks), admitted to the Neonatal Intensive Care Unit (NICU)

Exclusion Criteria:

* major congenital malformations or prenatal infections

Max Age: 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants with gestational age between 175-216 days (25-30 weeks), admitted to the Neonatal Intensive Care Unit (NICU) will be enrolled for this study. Saliva sample will be collected at least even seven days from the birth date and up to 40 weeks (286 days) of PMA or up to discharge if it occurs earlier
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Salivary biomarkers of oxidative stress to be associated with Bronchopulmonary dysplasia and/or Retinopathy of prematurity | From birth to 40 weeks of postmenstrual age
  The aim of the study will be to establish the structure and the relative amount over time of several peptides and proteins detectable in preterm saliva still pending for a precise characterization, with particular regard to enzymes with oxidative activity
Salivary biomarkers of proteolysis to be associated with Bronchopulmonary dysplasia and/or Retinopathy of prematurity | From birth to 40 weeks of postmenstrual age
  The aim of the study will be to establish the structure and the relative amount over time of several peptides and proteins detectable in preterm saliva still pending for a precise characterization, with particular regard to enzymes with proteolytic activity

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vento, MD, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No